CLINICAL TRIAL: NCT03342794
Title: Morphologic and Biometric Characteristics of Preexisting Posterior Capsule Defects in Congenital Cataracts During the First Year of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, Director, Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PCD_HZ
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Congenital Cataract
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- preexisting posterior capsule defects (Other): congenital cataracts with a preexisting posterior capsule defect
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — To diagnose the preexisting posterior capsule defects in congenital cataracts after the cataracts are removed by surgery and observe the characteristics

SUMMARY:
Few descriptive studies have focused on the anatomical parameters in patients with preexisting PCDs. The characteristics of cataract morphology and anatomical parameters in these patients remained unclear, when compared with CC patients with intact posterior capsule. We conduct the current study to compare the cataract morphology and preoperative parameters, including central corneal thickness, axial length, anterior chamber depth, lens thickness, corneal diameter, keratometry，dialated pupil diameter and intraocular pressure, between CC patients with preexisting PCDs and those with intact posterior capsule, and to explore potential risk factors for preexisting PCDs.

DETAILED DESCRIPTION:
This retrospective study reviewed infants (≤1 years old) with CC who were undergoing cataract extraction without IOL implantation at the Eye Hospital of Wenzhou Medical University, Hangzhou, China. CC patients with preexisting PCDs were placed in Study group, while CC patients with intact posterior capsule were included as controls.

The preexisting PCD was diagnosed if signs of a sharply bordered defect or white dots on the posterior capsule and/or in the anterior vitreous were detected. The intraoperative diagnosis of preexisting PCD was confirmed when the signs were observed after uneventful aspiration of the lens cortex. Patients who were incooperative to complete the preoperative examinations were excluded.

All CC patients were divided into two groups according to integrity of posterior capsule. Patients with a confirmed preexisting PCD were placed into the PCD group. Others with intact posterior capsule were in the control group. The preoperative data including sex, age at surgery, laterality of disease, and accompanying ocular anomalies were collected.

For all the CC patients, the preoperative examinations were completed under sedation. Central corneal thickness was obtained by a handheld ultrasonic pachymeter (PachPen, Accutome, US). Axial length, anterior chamber depth, lens thickness and length of vitreous cavity were measured via an immersion A-scan (Axis nano, Quantel Medical, French). An experienced examiner repeated the measurement 10 times and the mean value was included. The keratometry values and intraocular pressure were gained by a handheld keratometer (HandyRef-K, NIDEK, Japan) and a handheld tonometer (Icare, Vantaa, Finland), respectively. Diameter of cornea and dilated pupil (dilated by tropicamide 0.5% and phenylephrine hydrochloride 0.5%) was measured just before surgery.

All surgeries were performed by the same surgeon (Y.E.Z.) under general anesthesia. Bimanual irrigation/aspiration and 2-port 23G anterior vitrectomy were performed. Three ophthalmologists reviewed all surgical recordings. The integrity of posterior capsule was masked to them. Morphological characteristics of cataracts were documented before surgery. After removing opaque cortex and/or nucleus, the configuration of preexisting PCDs was described.

ELIGIBILITY:
Inclusion Criteria:

* congenital cataract

Exclusion Criteria:

* incooperative to complete the preoperative examinations

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
lens thickness measured by A-scan ultrasonography | 6 months
  lens thickness in congenital cataracts with either preexisting posterior capsule defects or intact posterior capsule will be measured by A-scan and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No